CLINICAL TRIAL: NCT06235203
Title: Neoadjuvant-Adjuvant Versus Adjuvant-Only Therapy Combined With Endoscopic Surgery in Advanced Recurrent Nasopharyngeal Carcinoma:A Multicenter Randomized Controlled Trial
Brief Title: Neoadjuvant vs Adjuvant in Locally Advanced Recurrent NPC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Shanghai 6th People's Hospital (Other); Changhai Hospital (Other); Fujian Medical University Union Hospital (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other); Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: adv-rNPC-RCT-Neo-V1
Record Dates: First submitted 2023-12-21; First posted 2024-01-31 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Recurrent Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Endoscopy; Neoadjuvant Therapy; toripalimab; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The control group (Active Comparator): Endoscopic surgery + adjuvant therapy
  Interventions: Procedure: endoscopic surgery; Drug: Adjuvant therapy in control group,Toripalimab Injection and Gemcitabine based therapy
- The experimental group (Experimental): Neoadjuvant therapy +endoscopic surgery + adjuvant therapy
  Interventions: Procedure: endoscopic surgery; Drug: Neoadjuvant therapy,Toripalimab Injection and Gemcitabine based therapy; Drug: Adjuvant therapy in experimental group,Toripalimab Injection and Gemcitabine based therapy

INTERVENTIONS:
Procedure: endoscopic surgery — The tumor was resected by endoscopic nasopharyngectomy.
Drug: Neoadjuvant therapy,Toripalimab Injection and Gemcitabine based therapy — Two courses of Toripalimab Injection and two courses of Toripalimab Injection and Gemcitabine based chemotherapy were given before endoscopic surgery.
  Arms: The experimental group
Drug: Adjuvant therapy in experimental group,Toripalimab Injection and Gemcitabine based therapy — Eight courses of Toripalimab Injection and two to four courses of chemotherapy, or until unacceptable side effects.
  Arms: The experimental group
Drug: Adjuvant therapy in control group,Toripalimab Injection and Gemcitabine based therapy — Ten courses of Toripalimab Injection and four to six courses of chemotherapy,or until unacceptable side effects.
  Arms: The control group

SUMMARY:
A multicenter randomized controlled study of surgery combined with neoadjuvant and adjuvant therapy for locally advanced recurrent nasopharyngeal carcinoma in comparison to surgery combined with adjuvant therapy

DETAILED DESCRIPTION:
Eligible patients are randomized into the control group and the experimental group.

Patients in the experimental group would be administrated 2 courses of neoadjuvant therapy before surgery.After endoscopic surgery, patients would continue to receive 2-4 courses of chemotherapy and 8 courses of immunotherapy.

Patients in the control group would firstly receive endoscopic surgery, followed by chemotherapy and immunotherapy. In total, 4 to 6 courses of chemotherapy and 10 courses of immunotherapy would be administrated.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically diagnosed with recurrent nasopharyngeal carcinoma;
2. Resectable disease staging rT2 (deep parapharyngeal space, or distance to the internal carotid ≤5mm) or rT3 (excluding the lesions confined to the basal wall of sphenoid sinus), rT4, according to AJCC 8th edition;
3. Cervical lymph node metastasis can be controlled locally;
4. Aged 18 to 75 years;
5. Informed consent forms signed to participate in the trial;
6. Without distant metastasis;
7. ≥6months from the accomplishment of radical radiation to recurrence
8. previously only 1 course of radiotherapy;
9. Sufficient organ function;
10. ECOG score 0-2 and can tolerate surgery,chemotherapy and immunotherapy.

Exclusion Criteria:

1. Participate in other interventional clinical trials;
2. Uncontrolled illnesses that interfere with the therapy;
3. Suffering from another or multiple malignancy within 5 years (excluding fully treated basal cell or skin squamous cell carcinoma, cervical carcinoma in situ, etc.);
4. Any contradiction to surgery;
5. With serious autoimmune disease;
6. The patient is currently using immunosuppressive agents or systemic hormone therapy to achieve immunosuppressive effects (dosage>10mg/day prednisone or other glucocorticoids), and continues to use them within 2 weeks before the first administration;
7. Severe allergic reactions to other monoclonal antibodies;
8. History of radioactive particle planting;
9. Vaccination with live vaccine within 4 weeks prior to initial administration or possibly during the study period;
10. Female patients who are at pregnancy or lactation;
11. Other situations that the researchers believe not suitable for enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
EFS | From randomization and any events(like:progression or toxic effects precluding surgery;inability to resect all gross disease; progression;surgical complications precluding initiation of adjuvant therapy; recurrence;death) up to 1 year
  Event free survival

SECONDARY OUTCOMES:
OS | Time interval of randomization and death of any cause, up to 5 years
  Overall Survival
DFS | From randomization to recurrence, metastasis or death, up to 1 year
  Disease free survival
LRFS | From randomization to local recurrence or death, up to 1 year
  Local recurrence free survival
DMFS | From randomization to distant metastasis or death, up to 1 year
  Distant metastasis free survival
pCR | Time point of pathological tumor evaluation after sugery, around 2 weeks after sugery
  pathologic complete response
ORR | Time point of imaging evaluation before treatment(or randomization) and before surgery,up to 1 year
  Objective response rate,Proportion of CR, PR in all patients.
DCR | Time point of imaging evaluation before treatment(or randomization) and before surgery,up to 1 year
  Disease Control Rate,Proportion of CR, PR and SD in all patients.
DoR | First date of response to the date of progression, up to 5 years
  Duration of response,the time from the first assessment of the tumour as CR or PR to the first assessment of PD or death from any cause (whichever event occurs first).
1-and 2-year PFS rate | one- and two-year
  one- and two-year progression free survival rate
1-and 2-year OS rate | one- and two-year
  one- and two-year overall survival rate

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Eye& ENT Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Fujian Medical University Union Hospital, Fuzhou
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning
  - Changhai Hospital, Shanghai
  - Shanghai Sixth People's Hospital, Shanghai
  - Shanghai Zhongshan Hospital, Shanghai
  - Shenzhen Second People's Hospital, Shenzhen

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR